CLINICAL TRIAL: NCT04328194
Title: Autotaxin (ATX) as a Marker for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mary Gamal Sudky, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: medicin
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — X-Rays; Ultrasonography, Mammary; Mammography; Magnetic Resonance Spectroscopy; Prothrombin Time

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): 80 patients with breast cancer
  Interventions: Diagnostic Test: Serum Autotaxin; Radiation: chest x-ray; Diagnostic Test: Breast ultrasound or mammography; Diagnostic Test: Histopathological examination of breast mass specimens; Radiation: Magnetic Resonance Imaging ( MRI) and Bone scan; Diagnostic Test: Peripheral haemogram; Diagnostic Test: Renal and liver functions; Diagnostic Test: Prothrombin time and concentration; Diagnostic Test: Cancer Antigen 15-3 (CA15-3).; Other: Full medical history; Other: Full clinical examination
- Control Group (Placebo Comparator): 20 healthy controls aged ( 19 to 69 years ) from healthy volunteers after informed consent.
  Interventions: Diagnostic Test: Serum Autotaxin; Diagnostic Test: Cancer Antigen 15-3 (CA15-3).; Other: Full medical history; Other: Full clinical examination

INTERVENTIONS:
Diagnostic Test: Serum Autotaxin — Marker
Radiation: chest x-ray — chest x- ray will be done for the study group
  Arms: Study Group
Diagnostic Test: Breast ultrasound or mammography — Breast ultrasound or mammography will be done for the study group to diagnosis of breast cancer
  Arms: Study Group
Diagnostic Test: Histopathological examination of breast mass specimens — by True cut or fine needle aspiration cytology
  Arms: Study Group
Radiation: Magnetic Resonance Imaging ( MRI) and Bone scan — will be done for the study group
  Arms: Study Group
Diagnostic Test: Peripheral haemogram — blood sample will be taken from the patients
  Arms: Study Group
Diagnostic Test: Renal and liver functions — to exclude any other morbidity
  Arms: Study Group
Diagnostic Test: Prothrombin time and concentration — blood sample will be taken from the patients
  Arms: Study Group
Diagnostic Test: Cancer Antigen 15-3 (CA15-3). — will be done for the 2 groups
Other: Full medical history — full medical history will be taken from all patients
Other: Full clinical examination — full clinical examination will be done for the patients

SUMMARY:
Breast cancer is the leading cause of cancer death in women worldwide. According to the GLOBOCAN 2018 worldwide estimates of cancer incidence and mortality, in 2018, about 2,088,849 new cases were diagnosed and approximately 626,679 women were predicted to die from the disease . It is the leading cause of cancer related mortality, representing15% of deaths per year worldwide .

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in females in Egypt. It accounts for 32 % of cancer in women . Breast cancer in Egypt carries an unfavorable prognosis with 29% mortality and 3.7:1 incidence to mortality ratio .

Despite the rising incidence of breast cancer, the survival rates have improved in recent years due to the deep research in biological behavior of breast cancer . Although the current 5-year survival for primary breast cancer is relatively high (ranging from 80% to 92% in different populations) survival rates decrease to less than 25% when the disease becomes metastatic .These data support the need to develop more efficient strategies for preventive, intervention, evaluation of therapy, and prediction of prognosis .

Autotaxin (ATX) is a glycoprotein encoded by the ENPP2 (Ectonucleotide Pyrophosphatase/Phosphodiesterase 2) gene located on chromosome 8. Identical to lysophospholipase D, ATX plays a role in the synthesis of the bioactive lipid mediator lysophosphatidate (LPA) from lysophosphatidylcholine (LPC) .

LPA acts through specific G protein-coupled receptors (GPCRs) to promote cellular proliferation, migration, and survival . ATX expression was also reported higher in poorly differentiated tumors and, in independent studies, is correlated with invasiveness of cancer cells suggesting a higher metastatic potential of ATX-expressing tumors . ATX is generated from platelets, endothelial cells, fibroblasts, and adipocytes and specifically, ATX from adipocytes has an impact on plasma LPA level . Thus, adipocytes could be an important origin of ATX in tumors. Breast cancer is a human cancer that has adipocyte-rich stroma. Adipose tissue comprises 56% of non-lactating breast tissue, and 35% of lactating breast tissue . ATX-LPA signaling has been reported to be involved in angiogenesis, tumor cell invasion, and migration in breast cancer .

Increased ATX expression has also been reported in various forms of cancer, such as glioblastoma, hepatocellular and thyroid carcinomas, pancreatic and hematological cancers. A large number of evidence indicate that ATX-LPA is associated with chemotherapy resistance of cancer, and in breast cancer, ATX can reverse cell apoptosis.

In a mouse model, α-bromomethylene phosphonate LPA (BrP-LPA), a dual ATX and pan-LPAR( Lysophosphatidic acid receptor ) inhibitor, inhibited migration and invasion of breast cancer cell lines and suppressed primary tumor and angiogenesis in a mouse xenograft study . Since tumor and stromal cells in breast cancer express ATX-LPA signaling-related proteins, inhibition of the ATX-LPA axis could be of therapeutic importance .Therefore, further study ATX as a tumor marker in breast cancer is required.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted on one hundred female individuals; 80 newly diagnosed breast cancer patients before any treatment or surgical intervention and 20 apparently normal female individuals.

Exclusion Criteria:

* Patients with any other type of malignant or benign tumors, renal failure, cardiovascular diseases and liver cirrhosis were excluded from our study.
* Past history of chemotherapy or surgical treatment of any malignancy.
* Inflammatory diseases (e.g.bronchitis) or autoimmune diseases (e.g.rheumatoid arthritis).

Ages: 19 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
To estimate the level of serum ATX as a diagnostic marker for breast cancer. | Baseline (before any treatment)
  blood sample will be taken from the patients for measure of serum ATX

SECONDARY OUTCOMES:
To establish a cut off for serum ATX as a marker for breast cancer | Baseline (before any treatment)
  blood sample will be taken from the patients for measure of serum ATX

REFERENCES:
- [Result] Boucharaba A, Serre CM, Gres S, Saulnier-Blache JS, Bordet JC, Guglielmi J, Clezardin P, Peyruchaud O. Platelet-derived lysophosphatidic acid supports the progression of osteolytic bone metastases in breast cancer. J Clin Invest. 2004 Dec;114(12):1714-25. doi: 10.1172/JCI22123. PMID 15599396
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Choi JW, Herr DR, Noguchi K, Yung YC, Lee CW, Mutoh T, Lin ME, Teo ST, Park KE, Mosley AN, Chun J. LPA receptors: subtypes and biological actions. Annu Rev Pharmacol Toxicol. 2010;50:157-86. doi: 10.1146/annurev.pharmtox.010909.105753. PMID 20055701
- [Result] Dusaulcy R, Rancoule C, Gres S, Wanecq E, Colom A, Guigne C, van Meeteren LA, Moolenaar WH, Valet P, Saulnier-Blache JS. Adipose-specific disruption of autotaxin enhances nutritional fattening and reduces plasma lysophosphatidic acid. J Lipid Res. 2011 Jun;52(6):1247-1255. doi: 10.1194/jlr.M014985. Epub 2011 Mar 18. PMID 21421848
- [Result] Ferry G, Tellier E, Try A, Gres S, Naime I, Simon MF, Rodriguez M, Boucher J, Tack I, Gesta S, Chomarat P, Dieu M, Raes M, Galizzi JP, Valet P, Boutin JA, Saulnier-Blache JS. Autotaxin is released from adipocytes, catalyzes lysophosphatidic acid synthesis, and activates preadipocyte proliferation. Up-regulated expression with adipocyte differentiation and obesity. J Biol Chem. 2003 May 16;278(20):18162-9. doi: 10.1074/jbc.M301158200. Epub 2003 Mar 17. PMID 12642576
- [Result] Hinestrosa MC, Dickersin K, Klein P, Mayer M, Noss K, Slamon D, Sledge G, Visco FM. Shaping the future of biomarker research in breast cancer to ensure clinical relevance. Nat Rev Cancer. 2007 Apr;7(4):309-15. doi: 10.1038/nrc2113. PMID 17384585
- [Result] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Result] Jansen S, Stefan C, Creemers JW, Waelkens E, Van Eynde A, Stalmans W, Bollen M. Proteolytic maturation and activation of autotaxin (NPP2), a secreted metastasis-enhancing lysophospholipase D. J Cell Sci. 2005 Jul 15;118(Pt 14):3081-9. doi: 10.1242/jcs.02438. Epub 2005 Jun 28. PMID 15985467
- [Result] Kazama S, Kitayama J, Aoki J, Mori K, Nagawa H. Immunohistochemical detection of autotaxin (ATX)/lysophospholipase D (lysoPLD) in submucosal invasive colorectal cancer. J Gastrointest Cancer. 2011 Dec;42(4):204-11. doi: 10.1007/s12029-010-9186-4. PMID 20623382
- [Result] Leblanc R, Peyruchaud O. New insights into the autotaxin/LPA axis in cancer development and metastasis. Exp Cell Res. 2015 May 1;333(2):183-189. doi: 10.1016/j.yexcr.2014.11.010. Epub 2014 Nov 25. PMID 25460336
- [Result] Lonning PE. Breast cancer prognostication and prediction: are we making progress? Ann Oncol. 2007 Sep;18 Suppl 8:viii3-7. doi: 10.1093/annonc/mdm260. PMID 17890212
- [Result] Mao Y, Keller ET, Garfield DH, Shen K, Wang J. Stromal cells in tumor microenvironment and breast cancer. Cancer Metastasis Rev. 2013 Jun;32(1-2):303-15. doi: 10.1007/s10555-012-9415-3. PMID 23114846
- [Result] Nikitopoulou I, Oikonomou N, Karouzakis E, Sevastou I, Nikolaidou-Katsaridou N, Zhao Z, Mersinias V, Armaka M, Xu Y, Masu M, Mills GB, Gay S, Kollias G, Aidinis V. Autotaxin expression from synovial fibroblasts is essential for the pathogenesis of modeled arthritis. J Exp Med. 2012 May 7;209(5):925-33. doi: 10.1084/jem.20112012. Epub 2012 Apr 9. PMID 22493518
- [Result] Ramsay DT, Kent JC, Hartmann RA, Hartmann PE. Anatomy of the lactating human breast redefined with ultrasound imaging. J Anat. 2005 Jun;206(6):525-34. doi: 10.1111/j.1469-7580.2005.00417.x. PMID 15960763
- [Result] Reis-Filho JS, Pusztai L. Gene expression profiling in breast cancer: classification, prognostication, and prediction. Lancet. 2011 Nov 19;378(9805):1812-23. doi: 10.1016/S0140-6736(11)61539-0. PMID 22098854
- [Result] Samadi N, Gaetano C, Goping IS, Brindley DN. Autotaxin protects MCF-7 breast cancer and MDA-MB-435 melanoma cells against Taxol-induced apoptosis. Oncogene. 2009 Feb 19;28(7):1028-39. doi: 10.1038/onc.2008.442. Epub 2008 Dec 15. PMID 19079345
- [Result] Teo K, Brunton VG. The role and therapeutic potential of the autotaxin-lysophosphatidate signalling axis in breast cancer. Biochem J. 2014 Oct 1;463(1):157-65. doi: 10.1042/BJ20140680. PMID 25195735
- [Result] van Meeteren LA, Moolenaar WH. Regulation and biological activities of the autotaxin-LPA axis. Prog Lipid Res. 2007 Mar;46(2):145-60. doi: 10.1016/j.plipres.2007.02.001. Epub 2007 Mar 16. PMID 17459484
- [Result] Vandeweyer E, Hertens D. Quantification of glands and fat in breast tissue: an experimental determination. Ann Anat. 2002 Mar;184(2):181-4. doi: 10.1016/S0940-9602(02)80016-4. PMID 11936199
- [Result] Windrichova J, Fuchsova R, Kucera R, Topolcan O, Fiala O, Finek J, Slipkova D, Karlikova M, Svobodova J. Testing of a Novel Cancer Metastatic Multiplex Panel for the Detection of Bone-metastatic Disease - a Pilot Study. Anticancer Res. 2016 Apr;36(4):1973-8. PMID 27069189
- [Result] Xia Q, Deng AM, Wu SS, Zheng M. Cholera toxin inhibits human hepatocarcinoma cell proliferation in vitro via suppressing ATX/LPA axis. Acta Pharmacol Sin. 2011 Aug;32(8):1055-62. doi: 10.1038/aps.2011.31. Epub 2011 Jul 18. PMID 21765444
- [Result] Shao Y, Yu Y, He Y, Chen Q, Liu H. Serum ATX as a novel biomarker for breast cancer. Medicine (Baltimore). 2019 Mar;98(13):e14973. doi: 10.1097/MD.0000000000014973. PMID 30921203
- [Result] Zhang S, Li L, Wang T, Bian L, Hu H, Xu C, Liu B, Liu Y, Cristofanilli M, Jiang Z. Real-time HER2 status detected on circulating tumor cells predicts different outcomes of anti-HER2 therapy in histologically HER2-positive metastatic breast cancer patients. BMC Cancer. 2016 Jul 25;16:526. doi: 10.1186/s12885-016-2578-5. PMID 27456503
- [Result] Zhang H, Xu X, Gajewiak J, Tsukahara R, Fujiwara Y, Liu J, Fells JI, Perygin D, Parrill AL, Tigyi G, Prestwich GD. Dual activity lysophosphatidic acid receptor pan-antagonist/autotaxin inhibitor reduces breast cancer cell migration in vitro and causes tumor regression in vivo. Cancer Res. 2009 Jul 1;69(13):5441-9. doi: 10.1158/0008-5472.CAN-09-0302. Epub 2009 Jun 9. PMID 19509223